CLINICAL TRIAL: NCT01716156
Title: A Phase II Randomized Clinical Trial to Study the Efficacy and Safety of MK-5172 in Combination With Ribavirin (RBV) in Subjects With Chronic Hepatitis C Virus Infection
Brief Title: A Study of Different Durations of Treatment With Grazoprevir (MK-5172) in Combination With Ribavirin in Participants With Chronic Hepatitis C (MK-5172-039)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5172-039; 2012-003340-72 (EudraCT Number)
Record Dates: First submitted 2012-10-25; First posted 2012-10-29 (Estimated); Results first posted 2016-03-04 (Estimated); Last update posted 2018-09-24 (Actual); Status verified 2018-08

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — grazoprevir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Grazoprevir 100 mg + RBV 12 Weeks (Experimental): Grazoprevir 100 mg tablet once per day by mouth for 12 weeks and RBV capsules twice per day by mouth at a total daily dose from 800 to 1400 mg based on participant weight for 12 weeks. Participants with detectable HCV RNA at TW4 received an additional 12 weeks of study therapy for a total of 24 weeks of treatment.
  Interventions: Drug: Grazoprevir; Drug: Ribavirin
- Grazoprevir 100 mg + RBV 24 Weeks (Experimental): Grazoprevir 100 mg tablet once per day by mouth for 24 weeks and RBV capsules twice per day by mouth at a total daily dose from 800 to 1400 mg based on participant weight for 24 weeks.
  Interventions: Drug: Grazoprevir; Drug: Ribavirin

INTERVENTIONS:
Drug: Grazoprevir — Grazoprevir, tablet, orally, 100 mg, once per day for 12 or 24 weeks, depending on Arm assignment
Drug: Ribavirin — Ribavirin capsules, orally, twice per day, at a total daily dose from 800 to 1400 mg based on participant weight
  Other Names: Rebetol™; RBV

SUMMARY:
This study will compare two different durations of treatment with grazoprevir (MK-5172) in combination with ribavirin (RBV) in treatment-naïve non-cirrhotic interferon-eligible interleukin 28b CC (IL28B CC) genotype participants with genotype 1 (GT1)-positive chronic hepatitis C (CHC). Participants will be randomized to receive 12 or 24 weeks of combination therapy.

ELIGIBILITY:
Inclusion Criteria:

* Chronic, compensated HCV GT 1 hepatitis C
* IL28B CC genotype
* Absence (no medical history or physical findings) of ascites, bleeding esophageal varices, hepatic encephalopathy, or other signs or symptoms of advanced liver disease, or cirrhosis
* No evidence of cirrhosis and hepatocellular carcinoma by biopsy or noninvasive tests (FibroScan and/or FibroTest)
* Agree to use two acceptable methods of birth control from at least 2 weeks prior to Day 1 and continue until at least 6 months after last dose of study drug, or longer if dictated by local regulations (for female subject who is of childbearing potential or male subject with female sexual partner who is of childbearing potential)

Exclusion Criteria:

* Non-GT 1 HCV infection, including a mixed GT infection (with a non-GT 1) or a non-typeable genotype
* Previous treatment with any interferon, RBV, approved or experimental direct acting antiviral(s), or other investigational therapies for HCV
* Human immunodeficiency virus (HIV) positive or known to be co-infected with hepatitis B virus
* Evidence of hepatocellular carcinoma (HCC) or under evaluation for HCC
* Currently participating or has participated in a study with an investigational compound within 30 days of signing informed consent and is not willing to refrain from participating in another study
* Diabetes and/or hypertension with clinically significant ocular examination findings
* Current moderate or severe depression or history of depression associated with hospitalization, electroconvulsive therapy, or severe disruption of daily functions, or suicidal or homicidal ideation and/or attempt, or history of severe psychiatric disorders
* Clinical diagnosis of substance abuse
* Current or history of seizure disorder, stroke, or transient ischemic attack
* Immunologically-mediated disease
* Chronic pulmonary disease
* Clinically significant cardiac abnormalities/dysfunction
* Active clinical gout within the last year
* Hemoglobinopathy or myelodysplastic syndromes
* History of organ transplants
* Poor venous access
* Indwelling venous catheter
* History of gastric surgery or malabsorption disorder
* Severe concurrent disease
* Evidence of active or suspected malignancy, or under evaluation for malignancy, or history of malignancy, within the last 5 years
* Pregnant, lactating, or expecting to conceive or donate eggs
* Male participant whose female partner is pregnant
* Member or a family member of the investigational study staff or sponsor staff directly involved with this study
* History of chronic hepatitis not caused by HCV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-01-18 (Actual); Primary Completion 2013-12-09 (Actual); Study Completion 2014-03-12 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Gane E, Ben Ari Z, Mollison L, Zuckerman E, Bruck R, Baruch Y, Howe AY, Wahl J, Bhanja S, Hwang P, Zhao Y, Robertson MN. Efficacy and safety of grazoprevir + ribavirin for 12 or 24 weeks in treatment-naive patients with hepatitis C virus genotype 1 infection. J Viral Hepat. 2016 Oct;23(10):789-97. doi: 10.1111/jvh.12552. Epub 2016 Jun 12. PMID 27291249

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 26 treatment-naive non-cirrhotic adult participants with hepatitis C virus (HCV) genotype 1 (GT1) were recruited in Australia, Israel, and New Zealand.
Pre-assignment Details: Allocation of participants to the 2 arms was stratified according to HCV GT1a vs. GT1b infection. Participants in the 12-week arm with detectable HCV ribonucleic acid (RNA) at Treatment Week (TW) 4 received 12 additional weeks of study treatment and are displayed in a separate treatment arm.
Groups:
- Grazoprevir 100 mg + RBV 12 Weeks Plus Extended: Grazoprevir 100 mg tablet once per day by mouth for 12 weeks and RBV capsules twice per day by mouth at a total daily dose from 800 to 1400 mg based on participant weight for 12 weeks. Participants with detectable HCV RNA at TW4 received an additional 12 weeks of study therapy for a total of 24 weeks of treatment.
Period: Overall Study
Arm/Group | Grazoprevir 100 mg + RBV 12 Weeks | Grazoprevir 100 mg + RBV 12 Weeks Plus Extended | Grazoprevir 100 mg + RBV 24 Weeks
Started | 9 | 4 | 13
Completed | 7 | 3 | 11
Not Completed | 2 | 1 | 2
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 2
Not completed — Lost to Follow-up | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Grazoprevir 100 mg + RBV 12 Weeks | Grazoprevir 100 mg + RBV 12 Weeks Plus Extended | Grazoprevir 100 mg + RBV 24 Weeks | Total
Number analyzed (Participants) | 9 | 4 | 13 | 26
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.1 (13.2) | 42.3 (7.4) | 42.8 (14.8) | 43.2 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 6 | 9
  Male | 7 | 3 | 7 | 17

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Sustained Virologic Response 12 Weeks After the End of All Study Therapy (SVR12)
Description: SVR12 was defined as HCV RNA <25 IU/mL 12 weeks after the end of all study therapy. HCV RNA was measured using the Roche COBAS™ Taqman™ HCV Test, v2.0® assay, which has a lower limit of quantification of 25 IU/mL and a limit of detection of 9.3 IU/mL.
Time Frame: Up to Week 36
Population: Per protocol population, as randomized. Per protocol population consists of all randomized participants receiving ≥1 dose of study therapy and no important protocol deviations.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Grazoprevir 100 mg + RBV 12 Weeks | Grazoprevir 100 mg + RBV 24 Weeks
Number analyzed (Participants) | 12 | 10
Percentage of participants | 58.3 [27.7 to 84.8] | 90.0 [55.5 to 99.7]

2. Primary Outcome: Percentage of Participants Experiencing at Least One Adverse Event (AE) on Study
Description: An adverse event is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An adverse event can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an adverse event. Data are presented according to actual treatment duration (12 weeks or 24 weeks) regardless of participants' initial arm assignment.
Time Frame: Fourteen days following last dose of study drug (up to 26 weeks)
Population: The All Participants as Treated (APaT) population included all randomized participants who received at least 1 dose of study therapy.
Measure: Number; unit: Percentage of participants
Groups:
- Grazoprevir 100 mg + RBV: up to 12 Weeks: The up to 12 weeks group consists of participants in the APaT population who only received 12 weeks of treatment and not those originally assigned to 12 weeks that went on to receive 24 total weeks of treatment.
- Grazoprevir 100 mg + RBV: Beyond 12 Weeks: The beyond 12 weeks group consists of participants in the APaT population who received 24 total weeks of treatment, regardless of original treatment regimen assignment.
Arm/Group | Grazoprevir 100 mg + RBV: up to 12 Weeks | Grazoprevir 100 mg + RBV: Beyond 12 Weeks
Number analyzed (Participants) | 11 | 15
Percentage of participants | 72.7 | 86.7

3. Primary Outcome: Percentage of Participants Discontinuing Study Therapy Due to an AE
Description: as for outcome 2
Time Frame: Up to 24 weeks
Population: The APaT population included all randomized participants who received at least 1 dose of study therapy.
Measure: Number; unit: Percentage of participants
Arm/Group | Grazoprevir 100 mg + RBV: up to 12 Weeks | Grazoprevir 100 mg + RBV: Beyond 12 Weeks
Number analyzed (Participants) | 11 | 15
Percentage of participants | 0 | 0

4. Secondary Outcome: Time to Achievement of First Undetectable HCV RNA
Description: The mean time (in days) to first achievement of undetectable HCV RNA was assessed using Kaplan-Meier plot and summary statistics. HCV RNA levels in plasma were measured using the Roche COBAS™ Taqman™ HCV Test, v2.0® assay on blood samples drawn from each participant at Week 2, Week 4, Week 12, and at end of treatment. The assay has a lower limit of quantification of 25 IU/mL and a limit of detection of 9.3 IU/mL. Undetectable HCV RNA was defined as below the limit of detection of 9.3 IU/mL.
Time Frame: Up to Week 24
Population: Full analysis set consists of all randomized participants receiving ≥1 dose of study therapy.
Measure: Mean (Standard Error); unit: Days
Groups:
- Grazoprevir 100 mg + RBV HCV GT1a: This group consisted of all participants with HCV GT1a infection pooled across treatment arms.
- Grazoprevir 100 mg + RBV HCV GT1non-a: This group consisted of all participants with HCV GT1non-a infection, pooled across treatment arms.
Arm/Group | Grazoprevir 100 mg + RBV HCV GT1a | Grazoprevir 100 mg + RBV HCV GT1non-a
Number analyzed (Participants) | 12 | 14
Days | 27.1 (2.5) | 19.7 (2.8)

5. Secondary Outcome: Percentage of Participants With Undetectable HCV RNA by Time Point
Description: HCV RNA levels in plasma were measured using the Roche COBAS™ Taqman™ HCV Test, v2.0® assay on blood samples drawn from each participant at Week 2, Week 4, Week 12, and at end of treatment (End of Treatment Response). The assay has a lower limit of quantification of 25 IU/mL and a limit of detection of 9.3 IU/mL. Undetectable HCV RNA was defined as below the limit of detection of 9.3 IU/mL.
Time Frame: From Week 2 through end of treatment (up to 24 weeks)
Population: Per protocol population, per assigned treatment duration. Per protocol population consists of all randomized participants receiving ≥1 dose of study therapy and no important protocol deviations.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Grazoprevir 100 mg + RBV 12 Weeks Extended: Grazoprevir 100 mg tablet once per day by mouth for 12 weeks and RBV capsules twice per day by mouth at a total daily dose from 800 to 1400 mg based on participant weight for 24 weeks. Participants with detectable HCV RNA at TW4 received an additional 12 weeks of study therapy for a total of 24 weeks of treatment.
Arm/Group | Grazoprevir 100 mg + RBV 12 Weeks | Grazoprevir 100 mg + RBV 12 Weeks Extended | Grazoprevir 100 mg + RBV 24 Weeks
Number analyzed (Participants) | 8 | 4 | 12
Percentage of participants
  Week 2 | 50.0 [15.7 to 84.3] | 0.0 [0.0 to 60.2] | 41.7 [15.2 to 72.3]
  Week 4; Grazoprevir 100 mg + RBV 24 Weeks, n=11 | 100.0 [63.1 to 100.0] | 0.0 [0.0 to 60.2] | 81.8 [48.2 to 97.7]
  Week 12; Grazoprevir 100 mg + RBV 24 Weeks, n=11 | 100.0 [63.1 to 100.0] | 75.0 [19.4 to 99.4] | 81.8 [48.2 to 97.7]
  End of all therapy | 100.0 [63.1 to 100.0] | 75.0 [19.4 to 99.4] | 91.7 [61.5 to 99.8]

6. Secondary Outcome: Percentage of Participants With HCV RNA <25 IU/mL by Time Point
Description: as for outcome 5
Time Frame: From Week 2 through end of treatment (up to 24 weeks)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Grazoprevir 100 mg + RBV 12 Weeks | Grazoprevir 100 mg + RBV 12 Weeks Extended | Grazoprevir 100 mg + RBV 24 Weeks
Number analyzed (Participants) | 8 | 4 | 12
Percentage of participants
  Week 2 | 100.0 [63.1 to 100.0] | 75.0 [19.4 to 99.4] | 100.0 [73.5 to 100.0]
  Week 4; Grazoprevir 100 mg + RBV 24 Weeks, n=11 | 100.0 [63.1 to 100.0] | 100.0 [39.8 to 100.0] | 100.0 [71.5 to 100.0]
  Week 12; Grazoprevir 100 mg + RBV 24 Weeks, n=11 | 100.0 [63.1 to 100.0] | 75.0 [19.4 to 99.4] | 90.9 [58.7 to 99.8]
  End of all therapy | 100.0 [63.1 to 100.0] | 75.0 [19.4 to 99.4] | 91.7 [61.5 to 99.8]

7. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 4 Weeks After Ending Study Therapy (SVR4)
Description: HCV RNA was measured using the Roche COBAS™ Taqman™ HCV Test, v2.0® assay, which has a lower limit of quantification of 25 IU/mL and a limit of detection of 9.3 IU/mL. SVR4 was defined as HCV RNA <25 IU/mL 4 weeks after the end of all study therapy.
Time Frame: Up to Week 28
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Grazoprevir 100 mg + RBV 12 Weeks | Grazoprevir 100 mg + RBV 12 Weeks Extended | Grazoprevir 100 mg + RBV 24 Weeks
Number analyzed (Participants) | 8 | 4 | 11
Percentage of participants | 87.5 [47.3 to 99.7] | 75.0 [19.4 to 99.4] | 90.9 [58.7 to 99.8]

8. Secondary Outcome: Percentage of Participants Achieving Sustained Virologic Response 24 Weeks After the End of Study Therapy (SVR 24)
Description: HCV RNA was measured using the Roche COBAS™ Taqman™ HCV Test, v2.0® assay, which has a lower limit of quantification of 25 IU/mL and a limit of detection of 9.3 IU/mL. SVR24 was defined as HCV RNA <25 IU/mL 24 weeks after the end of all study therapy.
Time Frame: Up to Week 48
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Grazoprevir 100 mg + RBV 12 Weeks | Grazoprevir 100 mg + RBV 12 Weeks Extended | Grazoprevir 100 mg + RBV 24 Weeks
Number analyzed (Participants) | 8 | 4 | 10
Percentage of participants | 62.5 [24.5 to 91.5] | 50.0 [6.8 to 93.2] | 80.0 [44.4 to 97.5]

ADVERSE EVENTS:
Time Frame: Up to 26 weeks (from first day of treatment, Day 1, through Day 14 of follow-up)
Description: APaT population consists of all randomized participants who received at least one dose of study treatment. Participants are included in the arm according to the duration of treatment received.
Arm/Group | Grazoprevir 100 mg + RBV: Beyond 12 Weeks | Grazoprevir 100 mg + RBV: up to 12 Weeks
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/11
Other Adverse Events (participants affected / at risk) | 13/15 | 8/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Grazoprevir 100 mg + RBV: Beyond 12 Weeks (N=15) | Grazoprevir 100 mg + RBV: up to 12 Weeks (N=11)
Hypertension (Vascular disorders) | 0 (0) | 1 (2)
Asthenia (General disorders) | 7 (7) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (2) | 0 (0)
Fatigue (General disorders) | 3 (3) | 1 (1)
Irritability (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Affective disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 4 (6) | 4 (10)
Eye inflammation (Eye disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (4) | 2 (3)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lip dry (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (3) | 2 (2)
Paraesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.